CLINICAL TRIAL: NCT03373123
Title: Radiomics-based Surrogate of Endoscopy (rEndosc) for Noninvasive Prediction of Esophageal Varices and Risk Stratification of Variceal Hemorrhage in Hepatitis B Virus-related Cirrhosis (CHESS1703)
Brief Title: Radiomics-based Surrogate of Endoscopy (rEndosc) (CHESS1703)
Acronym: rEndosc
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding issue
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Beijing YouAn Hospital (Other); Beijing 302 Hospital (Other); Shandong Provincial Hospital (Other Government); Beijing Friendship Hospital (Other); The Second Affiliated Hospital of Chongqing Medical University (Other); Chinese PLA General Hospital (Other); Peking University People's Hospital (Other); Xingtai People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaolong Qi, Director, Portal Hypertension Research, Institute of Hepatology, Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHESS1703
Record Dates: First submitted 2017-12-05; First posted 2017-12-14 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Esophageal Varices in Cirrhosis of the Liver
Keywords: Esophageal Varices; Variceal Hemorrhage; Endoscopy; Radiomics; Hepatitis B Virus
MeSH Terms: conditions — Esophageal and Gastric Varices; Hepatitis B | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm study (Experimental): Patients will receive CTA, Endoscopy, and rEndosc per protocol. Intervention: Procedure: Endoscopy
  Interventions: Procedure: Endoscopy; Procedure: CTA

INTERVENTIONS:
Procedure: Endoscopy — Endoscopy
Procedure: CTA — Radiomic features were extracted from CTA images.

SUMMARY:
Esophageal varices (EVs) resulting from portal hypertension are a prevalent complication of cirrhosis with a high mortality when variceal hemorrhage (VH) occurs. Screening endoscopy for EVs is recommended for all patients with cirrhosis, and prophylactic treatments are proposed for preventing VH, which may be financially onerous. Therefore, noninvasive tools for diagnosing EVs and risk stratifying VH in cirrhotic patients are needed to decrease the number of unnecessary invasive endoscopic examinations of low-risk patients and avoid unneeded prophylactic treatment. This is a prospective, multi-center diagnostic trial conducted at 9 high-volume liver centers in China designed to determine the diagnostic performance of radiomics-based surrogate (rEndosc) (investigational technology) by CT imaging for noninvasive prediction of EVs and risk stratification of VH in patients with hepatitis B virus-related cirrhosis using endoscopic examinations as reference standard.

DETAILED DESCRIPTION:
Esophageal varices (EVs) resulting from portal hypertension are a prevalent complication of cirrhosis with a high mortality when variceal hemorrhage (VH) occurs. Screening endoscopy for EVs is recommended for all patients with cirrhosis, and prophylactic treatments are proposed for preventing VH, which may be financially onerous. Therefore, noninvasive tools for diagnosing EVs and risk stratifying VH in cirrhotic patients are needed to decrease the number of unnecessary invasive endoscopic examinations of low-risk patients and avoid unneeded prophylactic treatment. This is a prospective, multi-center diagnostic trial conducted at 9 high-volume liver centers (Beijing YouAn Hospital, Capital Medical University; Nanfang Hospital, Southern Medical University; 302 Hospital of PLA; Shandong Provincial Hospital; Beijing Friendship Hospital, Capital Medical University; Chinese PLA General Hospital; Peking University People's Hospital; Xingtai People's Hospital) in China designed to determine the diagnostic performance of radiomics-based surrogate (rEndosc) (investigational technology) by CT imaging for noninvasive prediction of EVs and risk stratification of VH in patients with hepatitis B virus-related cirrhosis using endoscopic examinations as reference standard.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years;
* HBsAg positive;
* confirmed cirrhosis based on results of histologic examination of liver tissue or combined physical, laboratory, and radiologic findings, including a nodular surface, a coarse texture, and an enlarged caudate lobe of the liver on ultrasonography, CT, or MR imaging.

Exclusion Criteria:

* active alcohol abuse (less than 6 months of alcohol abstinence); portal thrombosis;
* history of treatments for portal hypertension (drug therapy, such as β-blocker, vasopressin) within 2 weeks;
* prior surgeries (such as splenectomy, partial splenic embolization/devascularization, transjugular intrahepatic portosystemic shunt);
* prior endoscopic therapies (such as endoscopic variceal ligation);
* previous variceal hemorrhage;
* acute-on-chronic (sub-acute) liver failure;
* malignant tumor (such as hepatocellular carcinoma);
* cirrhotic portal hypertension with isolated gastric varices or ectopic varices;
* inability to adhere to study procedures (such as heart failure, renal failure);
* pregnancy or unknown pregnancy status;
* no informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2018-12-18 (Estimated); Study Completion 2018-12-18 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of rEndosc for Esophageal Varices | 1 day
  Diagnostic accuracy of rEndosc to determine the presence or absence of esophageal varices when compared to endoscopic examination as the reference standard

SECONDARY OUTCOMES:
Diagnostic Accuracy of rEndosc for the Risk of Variceal Hemorrhage | 1 day
  Diagnostic accuracy of rEndosc to stratify risk of variceal hemorrhage when compared to endoscopic examination as the reference standard
Diagnostic Accuracy of rEndosc for Variceal Hemorrhage | 1 day
  Diagnostic accuracy of rEndosc to determine the presence or absence of variceal hemorrhage within 1-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Huiguo Ding, M.D., Principal Investigator — Beijing YouAn Hospital; Xiaolong Qi, M.D., Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (9):
- China (9):
  - 302 Hospital of PLA, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing YouAn Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Xingtai People's Hospital, Xingtai, Hebei
  - Shandong Provincial Hospital, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-Tsao G, Abraldes JG, Berzigotti A, Bosch J. Portal hypertensive bleeding in cirrhosis: Risk stratification, diagnosis, and management: 2016 practice guidance by the American Association for the study of liver diseases. Hepatology. 2017 Jan;65(1):310-335. doi: 10.1002/hep.28906. Epub 2016 Dec 1. No abstract available. PMID 27786365
- [Background] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Background] Gillies RJ, Kinahan PE, Hricak H. Radiomics: Images Are More than Pictures, They Are Data. Radiology. 2016 Feb;278(2):563-77. doi: 10.1148/radiol.2015151169. Epub 2015 Nov 18. PMID 26579733
- [Background] Segal E, Sirlin CB, Ooi C, Adler AS, Gollub J, Chen X, Chan BK, Matcuk GR, Barry CT, Chang HY, Kuo MD. Decoding global gene expression programs in liver cancer by noninvasive imaging. Nat Biotechnol. 2007 Jun;25(6):675-80. doi: 10.1038/nbt1306. Epub 2007 May 21. PMID 17515910
- [Background] Lambin P, Leijenaar RTH, Deist TM, Peerlings J, de Jong EEC, van Timmeren J, Sanduleanu S, Larue RTHM, Even AJG, Jochems A, van Wijk Y, Woodruff H, van Soest J, Lustberg T, Roelofs E, van Elmpt W, Dekker A, Mottaghy FM, Wildberger JE, Walsh S. Radiomics: the bridge between medical imaging and personalized medicine. Nat Rev Clin Oncol. 2017 Dec;14(12):749-762. doi: 10.1038/nrclinonc.2017.141. Epub 2017 Oct 4. PMID 28975929
- [Background] Huang YQ, Liang CH, He L, Tian J, Liang CS, Chen X, Ma ZL, Liu ZY. Development and Validation of a Radiomics Nomogram for Preoperative Prediction of Lymph Node Metastasis in Colorectal Cancer. J Clin Oncol. 2016 Jun 20;34(18):2157-64. doi: 10.1200/JCO.2015.65.9128. Epub 2016 May 2. PMID 27138577